CLINICAL TRIAL: NCT07120451
Title: Combination Therapy of Senaparib and Bevacizumab for First-line Maintenance Therapy in Newly Diagnosed Advanced Homologous Recombination Proficient Ovarian Cancer Based on Exosome Protein Marker: a Single Arm, Prospective Clinical Study
Brief Title: Combination Therapy of Senaparib and Bevacizumab for First-line Maintenance Therapy in Newly Diagnosed Advanced Homologous Recombination Proficient Ovarian Cancer Based on Exosome Protein Marker
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaohua Wu MD [zzhong], Director of Gynecological Oncology, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OC-SENABEV-HRP
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Advanced Ovarian Cancer
MeSH Terms: interventions — senaparib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Senaparib+Bevacizumab (Experimental): Participants will receive Senaparib and Bevacizumab in combination. Senaparib qd for 2 years and Bevacizumab q3w for 15 months.
  Interventions: Drug: Senaparib; Drug: Bevacizumab

INTERVENTIONS:
Drug: Senaparib — 100mg qd
Drug: Bevacizumab — 7.5mg/kg q3w

SUMMARY:
This study is a Prospective, Single-arm, Phase II clinical trial. The purpose of this study is to find out if taking combination therapy of Senaparib and Bevacizumab is safe and works well for people with first-line maintenance therapy in newly diagnosed advanced homologous recombination proficient ovarian cancer, and explore relevant biomarkers for evaluating the efficacy of maintenance therapy through exosome. Researchers will look at the Progression-Free Survival, Overall Survival, safety, and any side effects.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily joined this study, signed an informed consent form, had good compliance, and cooperated with follow-up;
2. Age range of 18 to 75 years old (calculated from the day of signing informed consent);
3. Patients with newly diagnosed epithelial ovarian cancer, fallopian tube cancer, and primary peritoneal cancer confirmed by histopathology;
4. FIGO stage III-IV, stage III subjects must have undergone one optimal tumor reduction surgery (first cell reduction surgery or intermittent cell reduction surgery). Participants in Phase IV studies must have undergone biopsy and/or first-time cytoreductive surgery or intermittent cytoreductive surgery; Can provide 10 pathological white films for subsequent research;
5. Tested as HRP
6. Achieving CR or PR after receiving platinum based treatment; CR refers to measurable and/or unmeasurable lesions without RECIST v1.1 criteria in imaging evaluation, and within the normal range of CA125. PR refers to the achievement of PR according to the RECIST v1.1 standard in imaging evaluation after chemotherapy, or the absence of measurable and/or unmeasurable lesions according to the RECIST v1.1 standard in imaging evaluation, with CA125 higher than the normal range and no sustained increase;
7. Before treatment, the CA125 test results must meet the following specific criteria:

If the first detection value is ≤ the upper limit of normal (ULN), the subjects can be randomly divided into groups without the need for a second sampling; If the first detection value is greater than ULN, a second evaluation must be conducted at least 7 days after the first detection. If the second evaluation value of the subject is higher than the first evaluation value by ≥ 15%, the subject is not eligible for selection; 8. Within 8-12 weeks of the last chemotherapy administration, participants must be enrolled and the trial medication must be started; 9. ECOG score: 0 to 1; 10. The main organ functions are normal and meet the following requirements (no blood components or cell growth factors are allowed to be used within 14 days before enrollment):

1. Blood routine examination: ① Hemoglobin (HB) ≥ 100g/L; ② Absolute neutrophil count (ANC) ≥ 1.5 × 10 ^ 9/L; ③ Platelet count (PLT) ≥ 1 × 10 ^ 11/L;
2. Blood biochemistry test: ① alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN (liver metastasis ≤ 5 × ULN); ② Serum total bilirubin (TBIL) ≤ 1.5 × ULN or direct bilirubin ≤ 1.0 × ULN; ③ Serum creatinine Cr ≤ 1.5 × ULN or creatinine clearance rate ≥ 60 ml/min;
3. Coagulation function test: activated partial thromboplastin time (APTT), international normalized ratio (INR), prothrombin time (PT) ≤ 1.5 × ULN; 11. Subjects with fertility are required to use at least one medically approved contraceptive measure (such as intrauterine device or condom) during the study treatment period and within 6 months after the last administration of the trial medication; And the serum HCG test result must be negative within 72 hours before the first administration; And it must be non lactating.

Exclusion Criteria:

1. Previous (within 5 years) or concurrent incurable malignant tumors, except for cured skin basal cell carcinoma, thyroid carcinoma, cervical carcinoma in situ, and breast cancer with no recurrence more than 3 years after the completion of radical surgery;
2. Have not previously used PARP inhibitors;
3. Those who are unable to swallow pills normally or have gastrointestinal dysfunction that may affect drug absorption, as determined by researchers;
4. Patients with a history of gastrointestinal perforation or major surgery within 4 weeks prior to the first use of medication; Patients with bleeding or bleeding events ≥ CTCAE grade 3, or with unhealed wounds, ulcers, or fractures;
5. Imaging (CT or MRI) shows tumor invasion of large blood vessels or unclear boundary with blood vessels;
6. Patients with poor blood pressure control (systolic blood pressure ≥ 150 mmHg and/or diastolic blood pressure ≥ 90 mmHg);
7. Urine routine shows that urine protein is ≥ 2+, and it is confirmed that the 24-hour urine protein content is ≥ 1.0 g;
8. Individuals who have experienced intestinal obstruction within the past 3 months;
9. Cancer ascites and pleural effusion with clinical symptoms that require puncture or drainage, or those who have received ascites or pleural effusion drainage within 2 months before the first trial medication;
10. Patients with abnormal coagulation function (INR>1.5 or prothrombin time (PT)>ULN+4 seconds), bleeding tendency, or undergoing thrombolytic or anticoagulant therapy are allowed to receive low-dose low-molecular-weight heparin or oral aspirin for anticoagulation prevention during the trial period;
11. Those who have used other drugs in clinical trials within the previous 4 weeks;
12. Prior to the first dose of the study drug, individuals who have received CYP3A4 potent inhibitors or CYP3A4 potent inducers (those with a half-life of ≥ 5 after elution from the first dose of the study drug can be enrolled) are not allowed to use CYP3A4 potent inhibitors or CYP3A4 potent inducers during the study period, as outlined in Appendix IV.
13. Participants may receive other systemic anti-tumor treatments during the study period;
14. Individuals known to be allergic to the excipients of Senaparib and Bevacizumab;
15. According to the researchers' assessment, there may be other factors that could lead to the forced termination of this study, such as other serious illnesses (including mental illnesses) requiring concurrent treatment, serious laboratory abnormalities, and family or social factors that could affect the safety of the subjects or the collection of data and samples.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
PFS | approximately 2 years
  Progression-free survival, according to RECIST v1.1

SECONDARY OUTCOMES:
OS | Up to 2 years
  Overall survival, according to RECIST v1.1
AEs | From the first drug administration to within 30 days for the last treatment dose
  Adverse Events, according to CTCAE V5.0 criteria, During the trial, the adverse event record form should be truthfully filled in, including the occurrence time, severity, correlation with study treatment, duration, measures taken and outcome of the adverse event.

OTHER OUTCOMES:
Detection of exosome related biomarkers | Up to 24 month
  Screening period, maintenance treatment for 1 month, 3 months, and disease progression will be tested separately

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Data is available per require after approved by ethics broad.